CLINICAL TRIAL: NCT03162406
Title: Effects of Vitamin D Supplementation During a Non-surgical Treatment of Generalized Chronic Periodontitis: A Randomized Double-blinded Placebo Controlled Clinical Trial
Brief Title: Effects of Vitamin D Supplementation During a Non-surgical Treatment of Generalized Chronic Periodontitis
Acronym: Protocol01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017/06JAN/013
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Generalized Chronic Periodontitis; Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D (Experimental): Procedure: SRP Dietary Supplement: Vitamin D3 Oral supplementation 25000 IU once per week for 6 months Other Name: Cholecalciferol
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): Procedure: SRP Dietary Supplement: Placebo Oral supplementation once per week for 6 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Oral supplementation 25000 IU once per week for 6 months
  Other Names: Cholecalciferol
  Arms: Vitamin D
Dietary Supplement: Placebo — Oral supplementation once per week for 6 months
  Other Names: Clear, slightly yellow, oily liquid with an orange odour
  Arms: Placebo

SUMMARY:
The subjects participating in the trial will be randomly allocated to either the group receiving the treatment under investigation (scaling and root planning (SRP) accompanied by administration of vitamin D) or to a group receiving standard treatment (SRP in conjunction with placebo) as the control. Random assignment of intervention will be done after subjects have been assessed for eligibility and recruited, but before the intervention to be studied begins. After randomization, the two groups of subjects will be followed in exactly the same way and the only differences between them will be the vitamin D/placebo that they will receive.

DETAILED DESCRIPTION:
It is likely that a chronically low intake of vitamin D and calcium may lead to a negative calcium balance, thus causing a secondary increase in calcium removal from bone, including the alveolar bone. Such bone loss may contribute to weakening of the tooth-attachment apparatus. In addition to its action on skeletal homeostasis, vitamin D, and, in particular, its hormonally active form, 1a,25-dihydroxyvitamin D, has anti-inflammatory and antimicrobial effects via modulation of inflammatory cytokine production by immune cells and stimulated secretion of peptides with antibacterial action by cells of the monocyte-macrophage lineage.These multiple actions of vitamin D are potentially appealing for the management of patients with periodontal disease, whose pathogenesis is based on chronic bacterial-driven inflammation.

Excess of vitamin D leads to a disturbance of the calcium in the body cycle. The symptoms experienced are: weakness, fatigue, headache, nausea, vomiting, diarrhea, polyuria, calciuria, dry mouth, nighttime urination, proteinuria, increased thirst, loss ofappetite, dizziness.

In case of high blood calcium level for a prolonged period, calcium deposits (tissue calcinosis) may occur in the soft tissues, including the kidneys where they cause calculations and calcium deposits in the nephrons, blood vessels, heart, lung and skin. These effects are reversible if the intoxication is detected in time.

ELIGIBILITY:
Inclusion Criteria:

* All subjects who are in good general health and were diagnosed with GChP (generalized chronic periodontitis) based on the current classification of the AmericanAcademy of Periodontology will be included:
* ≥ 30 years of age,
* at least 15 teeth (excluding third molars and teeth with advanced decay indicated for extraction),
* a minimum of 6 teeth with at least one site each with periodontal probing depth (PPD) and clinical attachment level (CAL) ≥ 5 mm,
* at least 30% of the sites with PPD and CAL ≥ 4 mm and bleeding on probing (BOP);
* Caucasians (defined as European and North African);
* subjects who present a 25(OH)D concentration < 30 ng/mL.

Exclusion Criteria:

* pregnancy
* breastfeeding
* current smoking and former smoking within the past 5 years-smoking status will be recorded as smoker (current) or non-smoker (never or former);
* systemic diseases that could affect the progression of periodontitis (e.g. diabetes, immunological disorders, osteoporosis);
* SRP in the previous 12 months;
* antibiotic therapy in the previous 6 months;
* long-term intake of anti-inflammatory medications;
* need for antibiotic pre-medication for routine dental therapy;
* any current ongoing immunological, neoplasia, endocrine, haematological, hepatic, renal, gastrointestinal, neurological, or psychiatric abnormalities or medical disease;
* subjects who used a UV light solarium or any type of vitamin D supplement within two months before the screening visit or planned to travel outside European countries during the study
* subjets under treatment with drugs that may interfere with vitamin D metabolism (e.g., phenobarbital, phenytoin, and glucocorticoids) and those with past or current history of granulomatosis, especially sarcoidosis, urinary lithiasis, and osteomalacia;
* subjects who present a 25(OH)D concentration > 30 ng/mL, serum creatinine >150 mmol/L and and albumin corrected serum calcium >2.65 mmol/L (corresponding to 10.6 mg/dL) at screening,
* any sensitivity or allergy to any of the products that will be used in the study or a history of drug and/or alcohol abuse.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects reaching ≤ 4 periodontal sites with PPD ≥ 5 mm | up to 6 months

SECONDARY OUTCOMES:
Number of sites with PPD ≥ 5 mm | up to 6 months
Number of sites with PPD ≥ 6 mm | up to 6 months
Number of sites with PPD ≥ 7 mm | up to 6 months
Reduction in the number of sites with PPD ≥ 5 mm | up to 6 months
Reduction in the number of sites with PPD ≥ 6 mm | up to 6 months
Reduction in the number of sites with PPD ≥ 7 mm | up to 6 months
Full-mouth PPD | up to 6 months
Full-mouth CAL | up to 6 months
Percentage of sites with BOP | up to 6 months
Percentage of sites with plaque accumulation | up to 6 months
Serum vitamin D concentration | 1 month before treatment and up to 6 months
Serum high-sensitivity C-reactive Protein (hs-CRP) | 1 month before treatment, at baseline, at 6 months
Serum high-density lipoprotein (HDL) cholesterol | 1 month before treatment, at baseline, at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Lasserre, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; Etienne Cavalier, PhD, Study Chair — Professor and Head of the Department of Clinical Chemistry, CHU Sart-Tilman Liège
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
It will be decided at the end of the study

REFERENCES:
- [Derived] Peric M, Maiter D, Cavalier E, Lasserre JF, Toma S. The Effects of 6-Month Vitamin D Supplementation during the Non-Surgical Treatment of Periodontitis in Vitamin-D-Deficient Patients: A Randomized Double-Blind Placebo-Controlled Study. Nutrients. 2020 Sep 25;12(10):2940. doi: 10.3390/nu12102940. PMID 32992785